CLINICAL TRIAL: NCT00201643
Title: A Randomized Double-Blinded Study Comparing the Impact of One Versus Two Courses of Antenatal Steroids on Neonatal Outcome
Brief Title: A Randomized Trial Comparing the Impact of One Versus Two Courses of Antenatal Steroids (ACS) on Neonatal Outcome
Acronym: ACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OBX0001; OBX0001 (Other: Obstetrix Medical Group)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Preterm Delivery
Keywords: Preterm Labor; Preterm delivery
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Betamethasone; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Test group (Active Comparator): Receive 2nd Course = Study drug (betamethasone or dexamethasone)
  Interventions: Drug: Betamethasone or Dexamethasone (2nd course of ACS)
- 2 - Control (Placebo Comparator): Placebo group = received placebo course
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Betamethasone or Dexamethasone (2nd course of ACS) — Course of Betamethasone or Dexamethasone
  Other Names: Beta; Dex
  Arms: 1 Test group
Drug: Placebo — Course of Placebo (NS)
  Other Names: Placebo, Normal Saline.
  Arms: 2 - Control

SUMMARY:
The hypothesis is that administration of two courses of antenatal corticosteroids, compared to one course, will show a 40% reduction in the incidence of composite neonatal morbidity in patients delivering prior to 34 weeks' gestation.

DETAILED DESCRIPTION:
This is a randomized double-blinded placebo-controlled trial. The objective of this study is to evaluate the impact of one versus two courses of antenatal steroids on the incidence of major neonatal morbidity including respiratory distress syndrome in patients delivering prior to 34 weeks' gestation in a randomized prospective fashion.

Preterm delivery occurs in approximately 10% of all deliveries in the United States. Preterm birth is the cause of 75% of neonatal mortality not mentioning the significantly increased morbidity from respiratory distress syndrome, intraventricular hemorrhage, necrotizing enterocolitis, and sepsis. Numerous studies have evaluated the safety and efficacy of antenatal corticosteroid (ACS) administration in threatened preterm labor.

National Institutes of Health (NIH) first consensus conference in 1994 evaluated the research in this field. Conclusions included the clear evidence that antenatal corticosteroids decrease the incidence of RDS in infants born at 29-34 weeks gestation, with a decrease in RDS severity for infants born at 24-28 weeks gestation and a decrease in the incidence of intraventricular hemorrhage in infants born at 24-28 weeks gestation without harm to mother or fetus. Their recommendation was to give a single course of corticosteroids to all pregnant women between 24 and 34 weeks gestation who are at risk of preterm delivery within 7 days.

Since the studies on the duration of the effects of antenatal corticosteroids in the fetus are not conclusive, many obstetricians repeat corticosteroids weekly or bi-weekly to patients continuing to be at risk for preterm delivery. Lacking scientific evidence, many investigators have performed retrospective analyses regarding the effects of single-course versus multiple-course antenatal corticosteroids.

The NIH consensus panel reconvened in 2000 and concluded that studies regarding repeated courses of corticosteroids are suggestive of possible benefits, especially in reduction of RDS, however, design flaws limit their validity.

The more recent publication from Caughey and Parer examined the literature for evidence regarding a dose response of the benefits and detriments of antenatal corticosteroids. Based on their complex mathematical analysis they recommend all fetus' between 24 and 34 weeks' gestation at risk for preterm delivery should be given a first course of ANC. If the risk of preterm delivery persists the next course should be given 2 weeks later, for a maximum of two courses. Consistent with all previous articles, the call for a well designed randomized, controlled trial is made.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 32 6/7 weeks gestation
* Singleton or twin gestation
* Received 1st course of betamethasone prior to 30 weeks' gestation
* Began 1st course of betamethasone at least 14 days prior to randomization
* Risk of delivery in next 7 days due to either maternal or fetal complication (e.g. preterm labor, severe preeclampsia, IUGR, etc.)
* Intact membranes

Exclusion Criteria:

* Known major fetal anomalies (eg: anencephaly, renal agenesis etc…)
* High order multiple gestation (triplets or higher)
* Cervical dilation > 5 cm
* Clinical chorioamnionitis prior to initiation of second course (two or more of the following; antepartum temperature > 38ºC (100.4ºF), uterine tenderness, foul smelling vaginal discharge or amniotic fluid, maternal tachycardia (>100beats/min), fetal tachycardia (>160 beats/min), or white blood cell count >20x109/L.define)
* Ruptured membranes prior to initiation of second course of betamethasone
* Already receiving corticosteroids for other conditions (e.g. Lupus, asthma)
* Maternal condition contraindicating the use of steroids (e.g. HIV, active Tuberculosis)
* Participation in conflicting study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 437 (Actual)
Dates: Start 2003-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Maurel, RN, MSN, CNS, Study Director — Obstetrix Medical Group, Inc.
Locations (22):
- United States (22):
  - Desert Good Samaritan Hospital, Mesa, Arizona
  - Banner Good Sammaritan Hospital, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of Sourthern California-Irvine Medical Center, Orange, California
  - Good Samaritan Hospital, San Jose, California
  - Swedish Medical Center, Denver, Colorado
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Skyridge Medical Center, Lonetree, Colorado
  - Mercy Medical Center, Des Moines, Iowa
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Saint Luke's Hospital, Kansas City, Kansas City, Missouri
  - Saint John's Regional Health Center, Springfield, Missouri
  - University Med. Ctr. of Southern Nevada, Las Vegas, Nevada
  - Sunrise Medical Center, Las Vegas, Nevada
  - Erlanger Medical Center, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Evergreen Hospital, Kirkland, Washington
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Background] Effect of corticosteroids for fetal maturation on perinatal outcomes. NIH Consens Statement. 1994 Feb 28-Mar 2;12(2):1-24. PMID 7728157
- [Background] Vermillion ST, Soper DE, Newman RB. Is betamethasone effective longer than 7 days after treatment? Obstet Gynecol. 2001 Apr;97(4):491-3. doi: 10.1016/s0029-7844(00)01178-9. PMID 11275015
- [Background] Antenatal corticosteroids revisited: repeat courses. NIH Consens Statement. 2000 Aug 17-18;17(2):1-18. PMID 11725806
- [Background] Guinn DA, Atkinson MW, Sullivan L, Lee M, MacGregor S, Parilla BV, Davies J, Hanlon-Lundberg K, Simpson L, Stone J, Wing D, Ogasawara K, Muraskas J. Single vs weekly courses of antenatal corticosteroids for women at risk of preterm delivery: A randomized controlled trial. JAMA. 2001 Oct 3;286(13):1581-7. doi: 10.1001/jama.286.13.1581. PMID 11585480
- [Background] Caughey AB, Parer JT. Recommendations for repeat courses of antenatal corticosteroids: a decision analysis. Am J Obstet Gynecol. 2002 Jun;186(6):1221-6; discussion 1226-9. doi: 10.1067/mob.2002.123742. PMID 12066102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women were recruited at 18 private (15) and university (3) medical centers from May 2003 through February 2008.
Pre-assignment Details: no washout, run-in or transition events occurred between enrollment and group assignment.
Groups:
- "Rescue" Course of Betamethasone or Dexamethasone: Receive 2nd "Rescue" Course = Study drug (betamethasone or dexamethasone. If Dexamethasone, administered 6 mg IM q 12 hours x 4 doses total. If Betamethasone was used, 2 doses of 12 mg of betamethasone was given intramuscularly (IM) 24 hours apart.
- Placebo (Normal Saline): Placebo consisted of quantity sufficient of Normal Saline with preservatives, Benzylalcohol and Benzylbenzoate.
  The research subject received 2 doses of pharmacy prepared placebo (2ml normal saline)to conceal administration of dexamethasone or if to conceal betamethasone, 2 doses of Placebo (2ml normal saline) given IM 24 hours apart.
Period: Overall Study
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Started | 223 | 214
Completed | 218 | 210
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 223 | 214 | 437
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 223 | 214 | 437
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6) | 29 (6) | 29 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 214 | 437
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 223 | 214 | 437

OUTCOME MEASURES:

1. Primary Outcome: Composite Neonatal Morbidity < 34 Weeks Gestation at Time of Birth.
Description: This outcome measured the total number of neonates with Composite Neonatal morbidity who delivered at < 34 weeks gestation. Composite Morbidity consisted of respiratory distress syndrome, bronchopulmonary dysplasia, severe intraventricular hemorrhage, periventricular leukomalacia, proven sepsis, necrotizing enterocolitis, or perinatal death
Time Frame: From birth to 28 days of life
Population: This was an intent to treat protocol. In patients delivering before 34 weeks we estimated that the sample size of at least 217 subjects in each arm would be needed to have 80% power to detect a 40% reduction in neonatal morbidity (to 16.8%).
Measure: Number; unit: participants
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 163 | 165
participants | 71 | 105
Statistical Analysis 1: Comparison: "Rescue" Course of Betamethasone or Dexamethasone vs Placebo (Normal Saline); Our Hypothesis was that administration of a rescue ACS would show a 40% reduction in incidence of composite neonatal morbity in patients delivering < 34 weeks. Sample size estimates based on composite morbidity of 28%. Each arm required 217 subjects to have 80% power to detect a 40% reduction to 16.8%(2-tailed,alpha =0.05)using comparison for proportions/groups(Fisher exact test) OR,95% CI & P values were determined using a repeated measure model where each twin is considered a repeat measure; Test type: Superiority or Other; p = 0.002, Fisher Exact — Analysis were also conducted in all randomized women with a known outcome & in randomized treatment group(modified intent to treat). Analysis of the primary outcome used a repeated measures approach where each baby was considered a repeated measure; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.27 to 0.75], Standard Error of Mean 0.1162

2. Secondary Outcome: Gestational Age at (@) Delivery
Description: Reported the average/mean Neonatal gestational age (GA) (reported in weeks of pregnancy) at the time of birth for both groups (ACS vs. Placebo).
Time Frame: gestational age at delivery in weeks of gestation
Population: Modified intent to treat
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 223 | 214
Weeks | 33.1 (3.1) | 33.0 (3.1)

3. Secondary Outcome: Neonatal Birth Weight Reported in Grams
Description: Measured mean Birth weights of Neonates in each arm as reported in grams on the birth record.
Time Frame: At time of Birth
Population: Intent to treat protocol
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 223 | 214
grams | 1905 (738) | 1920 (667)

4. Secondary Outcome: Interuterine Growth Restriction (IUGR) or Small for Gestational Age(SGA)in Babies Delivering at < 34 Weeks Gestation.
Description: Noted as the total number of Neonates delivering at < 34 weeks gestation for which their weights fell within the 10th percentile at time of birth.
Time Frame: Measured at birth.
Population: Intent to Treat
Measure: Number; unit: paticipants
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 162 | 161
paticipants | 25 | 20

5. Secondary Outcome: Neonatal Head Circumference Taken at Time of Birth.
Description: Reported as the average of all neonatal head circumferences (HC) taken at time of birth in each group.
Time Frame: Birth
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: centemeters (cm)
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 223 | 214
centemeters (cm) | 30.2 (3.0) | 30.0 (2.9)

6. Secondary Outcome: Number of Babies Who Required Ventilatory Support Within the First 28 Days of Life.
Description: The number of babies who required ventilatory support within the first 28 days of life. Equal to or great than 12 hours was considered one day.
Time Frame: birth to 28 days of life
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 267 | 273
participants | 70 | 95

7. Secondary Outcome: Number of Neonates Who Required Surfactant Therapy After Birth.
Description: The Number of neonates who required surfactant therapy within the first 28 days after birth.
Time Frame: Birth to 28 days of life
Population: ITT
Measure: Number; unit: participant
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 273 | 280
participant | 70 | 99

8. Secondary Outcome: Number of Neonates With Pneumothorax
Description: Total number of neonates with pneumothorax diagnosed postpartum.
Time Frame: birth to 28 days of life
Population: ITT
Measure: Number; unit: participants
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 275 | 281
participants | 4 | 4

9. Secondary Outcome: Maternal Infectious Morbidity.
Description: Total number of Mothers having Maternal infectious morbidity (e.g. endometritis & maternal sepsis) noted from birth through 28 days after birth
Time Frame: Up to 28 days after giving birth
Population: ITT
Measure: Number; unit: participants
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Number analyzed (Participants) | 223 | 214
participants | 8 | 10

ADVERSE EVENTS:
Time Frame: 4 years and (&) 9 months
Description: Evaluation of AEs occurred from randomization until 28days post delivery/discharge.
  The difference in reporting number(#)of participants at risk reflects the group for which the event relates to.e.g.: neonatal event N 289=test arm & 288=placebo
  * maternal event N 223=test arm & 214=placebo
  * maternal & neonatal 512= test arm & 502=placebo
Arm/Group | "Rescue" Course of Betamethasone or Dexamethasone | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 40/512 | 41/502
Other Adverse Events (participants affected / at risk) | 0/512 | 0/502
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | "Rescue" Course of Betamethasone or Dexamethasone (N=512) | Placebo (Normal Saline) (N=502)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Congenital Defect (Congenital, familial and genetic disorders) | 8/289 (10) | 12/288 (13) — to include: Congenital heart defects, hypospadias, inguinal hernia, hydrocele, dysmorphology, Cleft Lip, VATERS.
DIC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic Stenosis (Cardiac disorders) | 1/289 (1) | 1/288 (1)
Cardiac Dysfunction (Cardiac disorders) | 5/289 (5) | 2/288 (2) — Arrhythmias, cardiomyopathy, hypoperfusion
NEC (Gastrointestinal disorders) | 2/289 (2) | 5/288 (5)
Small Bowel Rotation (Gastrointestinal disorders) | 0/289 (0) | 1/288 (1)
Hyperbilirubenemia (Hepatobiliary disorders) | 2/289 (2) | 1/288 (1)
Hepatosplenomegally (Hepatobiliary disorders) | 0/289 (0) | 1/288 (1)
Wound infections (Infections and infestations) | 4/223 (4) | 3/214 (3)
Sepsis (Infections and infestations) | 2/289 (2) | 3/288 (3)
Mastitis (Infections and infestations) | 0/223 (0) | 1/214 (1)
Post delivery/C/S hemorrage (Injury, poisoning and procedural complications) | 4/223 (4) | 4/214 (4)
Spinal Headache (Injury, poisoning and procedural complications) | 1/223 (1) | 0/214 (0)
soft tissue rectal mass (Injury, poisoning and procedural complications) | 0/289 (0) | 1/288 (1)
Intraoperative Bladder Tear (Injury, poisoning and procedural complications) | 0/223 (0) | 1/214 (1)
PVL (Nervous system disorders) | 1/289 (1) | 0/288 (0)
Intraventicular Hemorrage (Grade III, IV) (Pregnancy, puerperium and perinatal conditions) | 2/289 (2) | 3/288 (3)
Perinatal fetal demise (Pregnancy, puerperium and perinatal conditions) | 2/289 (2) | 1/288 (1)
D & C for retained products (Surgical and medical procedures) | 1/223 (1) | 1/214 (1)
Abruption (Pregnancy, puerperium and perinatal conditions) | 0/223 (0) | 3/214 (3)
Apnea/respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1/289 (1) | 3/288 (3)
Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2/289 (2) | 0/288 (0) — Bronchiolitis, Pulmonary Interstitial Glycogenesis
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0/223 (0) | 1/214 (1)
Ruptured Appendix (Gastrointestinal disorders) | 0/223 (0) | 1/214 (1)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less